CLINICAL TRIAL: NCT04049929
Title: A Single-Arm, Open-Label, Multi-Center, Phase I Study of YY-20394 in Patients With Advanced Solid Tumors
Brief Title: A Phase I Study of YY-20394 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai YingLi Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YY-20394-003
Record Dates: First submitted 2019-07-21; First posted 2019-08-08 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-07

CONDITIONS: Advanced Solid Tumor
Keywords: YY-20394; Advanced solid tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YY-20394 (Experimental): YY-20394 tablets will be given daily for 28 days in 28-day cycles until there appears evidence of progressive disease, intolerable toxicity, or the subject discontinues from the study treatment for other reasons.
  Interventions: Drug: YY-20394

INTERVENTIONS:
Drug: YY-20394 — YY-20394 is a new type of PI3K-δ selective inhibitor which differs structurally from idelalisib and its analogs, showing high potency against PI3Kδ, but with markedly improved selectivity (>1,000-fold selectivity for PI3K-δ versus PI3Kγ). This higher selectivity for PI3Kδ may decrease the risk of serious infection seen with idelalisib and especially with duvelisib due to strong immune suppression.Preclinical evaluation has demonstrated improved efficacy and safety for YY-20394 compared to idelalisib.

SUMMARY:
Protocol YY-20394-003 is a phase I single arm, open label study. The primary objective is to assess the safety of YY-20394 in subjects with advanced solid tumor. The secondary objective is to determine the preliminary efficacy and pharmacokinetics (PK).

DETAILED DESCRIPTION:
In this clinical trials, patients will be dosed YY-20394 orally at 80mg per day until disease progression, unacceptable toxicity, or withdrawal from the study. A treatment cycle is defined as 28 days. Drug safety will be evaluated by NCI-CTC AE5.0 every week within 28 days after first dose and every 2 weeks in the following cycles. Efficacy will be assessed by RECIST1.1 after 2 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Males and/or females over age 18
2. Histologically or cytologically confirmed advanced solid tumors. Failure or lack of standard treatment.
3. Eastern Cooperative Oncology Group performance status of 0 to 2
4. Life expectancy of at least 3 months
5. At least one measurable lesion according to RECIST1.1.
6. Acceptable hematologic status:

   Absolute neutrophil count(ANC)≥1.5×10^9/L; Platelet count(PLT)≥75×10^9/L; Hemoglobin(Hb)≥80 g/L; Total bilirubin(TBIL)≤1.5×Upper limit of normal value(ULN); Alanine aminotransferase(ALT)≤1.5×ULN; Aspartate aminotransferase(AST)≤1.5×ULN; Creatinine(Cr)≤1.5×ULN; Left Ventricular Ejection Fractions(LVEF)≥50%； QTcF：male<450 ms,female<470 ms
7. Accept to use proper contraceptives throughout the study period and within 6 months after the last dose.
8. Ability to respect the protocol approved by investigator.
9. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Previously treated with PI3Kδ inhibitors and cause disease progression (removed from the study because of intolerance is not included).
2. Any anti-tumor treatment, within 4 weeks prior to study entry, such as chemotherapy, radiotherapy and immunotherapy. Nitrosoureas or mitomycin C within 6 weeks prior to study entry. Oral drug of fluorouracil or small molecular targeted drugs 2 weeks prior to study entry.
3. Any other investigational agents within 4 weeks prior to study entry.
4. Any surgery on main organ (needle biopsy not included) or serious injury within 4 weeks prior to study entry. Selective operation is required during the study period.
5. Adverse events of previous anti-cancer treatment have not recovered to CTCAE v5.0 ≤1.
6. There are third interstitial effusions (such as massive pleural effusion and ascites) which can not be controlled by drainage or other methods.
7. The dosage of steroid hormone (prednisone equivalent) was greater than 20mg/day, and lasted for more than 14 days.
8. Medical history of difficulty in swallowing, malabsorption, or other chronic gastrointestinal disease, or conditions that may hamper compliance and/or absorption of the tested drug.
9. During the study period, drugs that may prolong the QT (such as anti arrhythmic drugs) could not be interrupted.
10. Patients with central nervous system (CNS) matastasis or meningeal metastasis with clinical symptoms, or there are evidences of CNS matastasis or meningeal metastasis uncontrolled approved by investigators.
11. Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy(such as pneumonia).
12. Active hepatitis b (HBV titers>1000 copies/ml or 200IU/ml), prophylactic antiviral therapies other than interferon are allowed. Patients with Hepatitis C virus (hepatitis C antibody test positive).
13. History of immunodeficiency, including HIV positive test, other acquired or congenital immunodeficiency disorders, organ transplantation or allogeneic bone marrow transplantation.
14. Has suffered from any heart disease within 6 months prior to study entry, including: (1) angina pectoris; (2) medicated or clinically significant arrhythmia; (3) myocardial infarction; (4) heart failure; (5) any other heart disease judged by the researchers not suitable for the test.
15. The baseline pregnancy test was positive in pregnant women, lactating women or fertile women.
16. According to the judgement of the investigator, there are concomitant diseases that seriously endanger the safety of patients or affect the completion of the study (such as severe hypertension, diabetes, thyroid diseases, etc.
17. Patients suffering from other primary malignant tumors in the past 5 years. Patients with curable local tumors (such as basal or squamous cell carcinoma, superficial bladder cancer, carcinoma in situ of the cervix or of the breast) could be enrolled after completely cured.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Adverse events evaluated by NCI CTCAE v5.0 | with in 2 years after the first dose
  Incidence of adverse events of YY-20394

SECONDARY OUTCOMES:
Objective response rate | with in 56 days after the first dose
  Response will be determined by Response evaluation criteria in solid tumours; v1.1
Disease control rate | with in 56 days after the first dose
  DCR will be determined by Response evaluation criteria in solid tumours v1.1
Maximum concentration (Cmax) | 10 mins pre-dose in D1, D7, D14; 0.5, 1, 2, 4, 6, 8, 24 hours after the first dose
  One of Pharmacokinetic (PK) parameters.
Time to maximum concentration (Tmax) | 10 mins pre-dose in D1, D7, D14; 0.5, 1, 2, 4, 6, 8, 24 hours after the first dose
  One of Pharmacokinetic (PK) parameters.
Minimum concentration(Cmin) | 10 mins pre-dose in D1, D7, D14; 0.5, 1, 2, 4, 6, 8, 24 hours after the first dose
  One of Pharmacokinetic (PK) parameters.
Area under the curve (AUC) | 10 mins pre-dose in D1, D7, D14; 0.5, 1, 2, 4, 6, 8, 24 hours after the first dose
  One of Pharmacokinetic (PK) parameters.
Half-life (t1/2) | 10 mins pre-dose in D1, D7, D14; 0.5, 1, 2, 4, 6, 8, 24 hours after the first dose
  One of Pharmacokinetic (PK) parameters.
Clearance (CL) | 10 mins pre-dose in D1, D7, D14; 0.5, 1, 2, 4, 6, 8, 24 hours after the first dose
  One of Pharmacokinetic (PK) parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Hanying Bao, PhD, Study Director — Shanghai YingLi Pharmaceutical Co. Ltd.
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Eisenreich A, Rauch U. PI3K inhibitors in cardiovascular disease. Cardiovasc Ther. 2011 Feb;29(1):29-36. doi: 10.1111/j.1755-5922.2010.00206.x. PMID 20626398
- [Result] Samuels Y, Wang Z, Bardelli A, Silliman N, Ptak J, Szabo S, Yan H, Gazdar A, Powell SM, Riggins GJ, Willson JK, Markowitz S, Kinzler KW, Vogelstein B, Velculescu VE. High frequency of mutations of the PIK3CA gene in human cancers. Science. 2004 Apr 23;304(5670):554. doi: 10.1126/science.1096502. Epub 2004 Mar 11. No abstract available. PMID 15016963
- [Result] Yuan TL, Cantley LC. PI3K pathway alterations in cancer: variations on a theme. Oncogene. 2008 Sep 18;27(41):5497-510. doi: 10.1038/onc.2008.245. PMID 18794884
- [Result] Kong D, Yamori T. Phosphatidylinositol 3-kinase inhibitors: promising drug candidates for cancer therapy. Cancer Sci. 2008 Sep;99(9):1734-40. doi: 10.1111/j.1349-7006.2008.00891.x. Epub 2008 Jul 4. PMID 18616528
- [Result] Brown JR, Byrd JC, Coutre SE, Benson DM, Flinn IW, Wagner-Johnston ND, Spurgeon SE, Kahl BS, Bello C, Webb HK, Johnson DM, Peterman S, Li D, Jahn TM, Lannutti BJ, Ulrich RG, Yu AS, Miller LL, Furman RR. Idelalisib, an inhibitor of phosphatidylinositol 3-kinase p110delta, for relapsed/refractory chronic lymphocytic leukemia. Blood. 2014 May 29;123(22):3390-7. doi: 10.1182/blood-2013-11-535047. Epub 2014 Mar 10. PMID 24615777
- [Result] Flinn IW, Kahl BS, Leonard JP, Furman RR, Brown JR, Byrd JC, Wagner-Johnston ND, Coutre SE, Benson DM, Peterman S, Cho Y, Webb HK, Johnson DM, Yu AS, Ulrich RG, Godfrey WR, Miller LL, Spurgeon SE. Idelalisib, a selective inhibitor of phosphatidylinositol 3-kinase-delta, as therapy for previously treated indolent non-Hodgkin lymphoma. Blood. 2014 May 29;123(22):3406-13. doi: 10.1182/blood-2013-11-538546. Epub 2014 Mar 10. PMID 24615776
- [Result] Gopal AK, Kahl BS, de Vos S, Wagner-Johnston ND, Schuster SJ, Jurczak WJ, Flinn IW, Flowers CR, Martin P, Viardot A, Blum KA, Goy AH, Davies AJ, Zinzani PL, Dreyling M, Johnson D, Miller LL, Holes L, Li D, Dansey RD, Godfrey WR, Salles GA. PI3Kdelta inhibition by idelalisib in patients with relapsed indolent lymphoma. N Engl J Med. 2014 Mar 13;370(11):1008-18. doi: 10.1056/NEJMoa1314583. Epub 2014 Jan 22. PMID 24450858
- [Result] Furman RR, Sharman JP, Coutre SE, Cheson BD, Pagel JM, Hillmen P, Barrientos JC, Zelenetz AD, Kipps TJ, Flinn I, Ghia P, Eradat H, Ervin T, Lamanna N, Coiffier B, Pettitt AR, Ma S, Stilgenbauer S, Cramer P, Aiello M, Johnson DM, Miller LL, Li D, Jahn TM, Dansey RD, Hallek M, O'Brien SM. Idelalisib and rituximab in relapsed chronic lymphocytic leukemia. N Engl J Med. 2014 Mar 13;370(11):997-1007. doi: 10.1056/NEJMoa1315226. Epub 2014 Jan 22. PMID 24450857
- See also: Diagnosis, prognosis and treatment of chronic lymphoblastic leukemia (CLL) — http://www.wanfangdata.com.cn/details/detail.do?_type=conference&id=7408347
- See also: Correlation of P13K-Akt Signal Pathway to Apoptosis of Tumor Cells — http://www.wanfangdata.com.cn/details/detail.do?_type=perio&id=ez200803022